CLINICAL TRIAL: NCT04979650
Title: Corticosteroid Pulse Therapy Effects on MRI Asymptomatic Gadolinium-enhancing Lesions Conversion to a Non-enhancing Black Hole With or Without Treatment in MS Clinic of Booalisina Hospital Sari 2021-2023
Brief Title: Corticosteroid Effects on Asymptomatic Gadolinium-enhancing Lesions in Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mazandaran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Seyed Mohammad Baghbanian, Seyed Mohammad Baghbanian, Mazandaran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 978445
Record Dates: First submitted 2021-07-02; First posted 2021-07-28 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2021-07

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting; Magnetic Resonance Imaging; Methylprednisolone
Keywords: Multiple sclerosis; Methylprednisolone Pulse therapy; Asymptomatic enhancing lesions; Chronic black hole
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Methylprednisolone Hemisuccinate; Exercise; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The intervention group (Active Comparator): The intervention group will receive 1 gram of methylprednisolone succinate within 500 ccs of normal saline within 5 hours.
  Interventions: Drug: Methylprednisolone succinate; Drug: Normal saline
- The control group (Placebo Comparator): The control group will receive 500 g of normal saline without methylprednisolone succinate.
  Interventions: Drug: Methylprednisolone succinate; Drug: Normal saline

INTERVENTIONS:
Drug: Methylprednisolone succinate — 1 gram of methylprednisolone succinate within 500 ccs of normal saline
  Other Names: Active
Drug: Normal saline — 500 g of normal saline without methylprednisolone succinate
  Other Names: Placebo

SUMMARY:
to determine the rate of asymptomatic gadolinium-enhancing lesions conversion to the non-enhancing black hole (neBHs) with or without corticosteroid pulse therapy in patients with RRMS, and to analyze if treatment of asymptomatic gadolinium enhancement lesions has any effect on the expanded disability status scale. The study is performed in the MS clinic of Bu Ali Sina Hospital in Sari and Mazandaran University of Medical Sciences. 104 recurrent MS patients are admitted based on the admission criteria. They are divided into two groups of intervention and control based on a simple randomization block. The intervention group received 1 gram of methylprednisolone in 500 ccs of normal saline for 5 days and the control group received only 500 ccs of serum. After 6 months, a new MRI is taken from the patients and the possibility of asymptomatic active plaque conversion with or without intervention is compared in the two groups, as well as the amount of EDSS in the two groups. They do not know whether the patient is in the control group or the intervention.

DETAILED DESCRIPTION:
Investigators perform a study on 104 consecutive patients with a diagnosis of RR-MS. Participants will be selected for the study if they meet all of the following inclusion criteria: (1) a baseline MRI scan with at least one CEL on contrast-enhanced T1-weighted images (performed either at the time of the diagnosis or during the routine MRI monitoring of the disease) and (2) a follow-up MRI scan performed at least 6 months later in the same hospital site. Participants were then divided into two groups by block randomization (the Block size will be 4): (1) participants with asymptomatic CELs, treated with a single cycle of high-dose IVMP after baseline MRI (group A) and (2) participants with asymptomatic CELs for clinical relapse and, therefore, not exposed to IVMP after baseline MRI (group B).

1. Microsoft Excel software will be used for block randomization with a group of 4.
2. Number the participants from 1 to 102.
3. In a group of 2, the possible combinations of blocks are:(A=Group1 and B=Group2)

1. ABBA 2. ABAB 3. BBAA 4. ABAB 5. BAAB 6. BABA

To determine the sample size for this study we used the result of Maria Di Gregorio and et al.

This study will be double-blind patients and radiologist clinicians unaware of types of interventions.

MRI examinations were performed with a 1.5 T magnet (General Electric Medical Systems, Milwaukee, WI, USA) with a standard head coil. The MRI protocol used in our Neuroradiology Section included the following sequences: (1) a T2-weighted-fluid-attenuated inversion recovery (FLAIR) sequence with an inversion time (TI) of 2400 ms, an echo time (TE) of 120 ms, and a repetition time (TR) of 8000 ms; (2) a T2-weighted fast spin-echo (FSE) sequence with a TE of 90 ms and a TR of 6600 ms; and (3) a spin-echo (SE) sequence for T1-weighted images with a TR of 500 ms and a TE of 20 ms Post-contrast images were obtained with a scan delay of 5 min after the injection of gadoterate (Dotarem, Guerbet group, Roissy, France) at 0.2 mmol/kg. 3-mm thick contiguous slices were obtained.

In the baseline MRI, the following characteristics of CELs were recorded: (1) number; (2) maximum diameter (≤ or > 5 mm); (3) pattern of enhancement (homogeneous or ring enhancement); (4) hypointensity as compared to normal-appearing surrounding white matter in baseline T1-weighted images acute black hole (aBH); and (5) the fact of being symptomatic, as established by an experienced neurologist (MDG) on the basis of CELs' localization and clinical characteristics of the concomitant relapse. The follow-up MRI was performed with the same 1.5 T magnet and using the same MRI protocol. At the follow-up MRI, the presence of persistent black holes (pBHs) was recorded. Specifically, pBHs were defined as non-enhancing T1 lesions hypointense with respect to the surrounding normal-appearing white matter and concordant with hyperintense T2 lesions [10]. Three investigators (MDG, AP, and GR) in agreement with a senior experienced neuro-radiologist (PF) revised baseline CELs and follow-up pBHs' characteristics. The three investigators and the neuroradiologist were blinded to the exposure of the patients to IVMP treatment

ELIGIBILITY:
Inclusion Criteria:

* All patients with a diagnosis of RR-MS
* with a baseline MRI scan with at least one asymptomatic CEL on contrast-enhanced T1-weighted images

Exclusion Criteria:

* Pulse therapy 3 months ago,
* More than 6 months ago slowly progressive disease
* Systemic infections, including fungal infection
* Uncontrolled hypertension
* With known hypersensitivity to the steroid preparation

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2021-05-22 (Actual); Primary Completion 2023-12-28 (Actual); Study Completion 2023-12-29 (Actual)

PRIMARY OUTCOMES:
Number of black hole | After 6 months
  NeBH (to non-enhancing black hole) was defined as an area of unequivocal low signal intensity compared with normal-appearing white matter that did not show contrast uptake and was concordant with a hyperintense lesion seen on T2-weighted imaging.They have also been defined as T1-hypointensities persisting for more than 6 months after their appearance
Expanded disability status scale | After 6 months
  The EDSS quantifies disability in eight functional systems: pyramidal, cerebellar, brainstem, sensory, bowel and bladder, visual, cerebral, and other. It ranges from 1.0 to 4.5 for people affected with MS who are fully ambulatory, and from 5.0 to 9.5 for people with MS with impaired ambulation. The maximum grade, 10.0, represents death due to MS

CONTACTS AND LOCATIONS:
Overall Officials: Seyed Mohammad Baghbanian, Dr., Principal Investigator — Mazandaran University of Medical Sciences
Locations (1):
- Mazandaran University of medical sciences, Sari, Mazandaran, Iran

IPD SHARING:
Plan to Share IPD: Yes
All data is potentially shareable after unidentified individuals.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The access period starts 6 months after the results are published.
Access Criteria: It will be available only to researchers working in academic and scientific institutions.